CLINICAL TRIAL: NCT00099931
Title: Efficacy and Safety of Vildagliptin in Combination With Insulin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2311
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
Many people with type 2 diabetes cannot maintain their target blood glucose levels on a single therapy. The purpose of this study is to assess the safety and effectiveness of vildagliptin, an unapproved drug, in lowering overall blood glucose levels when added to insulin in people with type 2 diabetes who are not at target blood glucose levels on insulin alone.

ELIGIBILITY:
Inclusion Criteria:

* Blood glucose criteria must be met
* On a stable dose of insulin as defined by the protocol
* Body mass inde (BMI) in the range 22-45

Exclusion Criteria:

* Type 1 diabetes
* Pregnancy or lactation
* Evidence of serious diabetic complications
* Evidence of serious cardiovascular complications
* Laboratory value abnormalities as defined by the protocol
* Other protocol defined exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2004-05; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose at 24 weeks
Adverse event profile after 24 weeks of treatment
Change from baseline in mean daily insulin dose at 24 weeks
Change from baseline in mean daily number of insulin injections at 24 weeks
Patients with endpoint <7% after 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Investigative Sites, Germany

REFERENCES:
- [Derived] Fonseca V, Schweizer A, Albrecht D, Baron MA, Chang I, Dejager S. Addition of vildagliptin to insulin improves glycaemic control in type 2 diabetes. Diabetologia. 2007 Jun;50(6):1148-55. doi: 10.1007/s00125-007-0633-0. Epub 2007 Mar 27. PMID 17387446